CLINICAL TRIAL: NCT02108158
Title: A Randomized, Evaluator-blinded, Comparative Study to Evaluate the Efficacy and Safety of Different Injection Volumes of Botulinum Toxin Type A, Azzalure, in the Glabellar Lines
Brief Title: A Safety and Efficacy Study of Different Injections Volumes of Botulinum Toxin Type A, Azzalure, in the Glabellar Lines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05PF1311; 2013-004646-42 (EudraCT Number)
Record Dates: First submitted 2014-03-05; First posted 2014-04-09 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2015-08

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — abobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azzalure 10 Speywood units/injection (Experimental): Azzalure (botulinum toxin type A), powder for solution for injection, Total dose 50 s.U (5 x 10s.U)
  Interventions: Drug: Azzalure
- Azzalure, 10 Speywood units/injection (Active Comparator): Azzalure (botulinum toxin type A), powder for solution for injection, Total dose 50 s.U (5 x 10s.U)
  Interventions: Drug: Azzalure

INTERVENTIONS:
Drug: Azzalure
  Other Names: botulinum toxin type A

SUMMARY:
A randomized, evaluator-blinded, comparative, study to evaluate the efficacy and safety of different injection volumes of botulinum toxin type A, Azzalure, in the glabellar lines.

DETAILED DESCRIPTION:
Clarification regarding injection volumes for the different study groups:

Subjects will be randomized to Group A or Group B (1:1).

* Group A: 0,63ml NaCl will be used to reconstitute toxin in the vial. 0,05mL will be injected (equal to a dose of 10s.U.)
* Group B: 1,25ml NaCl will be used to reconstitute toxin in the vial. 0,1 mL will be injected (equal to a dose of 10s.U.).

The two different reconstitution volumes (each containing a dose of 10s.U. botulinum toxin A) will be compared as described under objectives.

ELIGIBILITY:
Key Inclusion Criteria:

* Women, 18 to 64 years of age
* Subjects seeking treatment for moderate to severe glabellar lines when the severity of these lines has an important psychological impact on the subject, as determined by the investigator.

Key Exclusion Criteria:

* Subjects previously treated with any botulinum toxin product.
* Pregnant or breast feeding women or women intending to get pregnant in the next 12 months.
* Subjects with signs and symptoms of eyelid or brow ptosis or signs of compensatory frontalis muscle activity, as judged by the investigator.
* Subjects with clinical or subclinical neuromuscular junctional disorders (e.g. myasthenia gravis, Lambert Eaton syndrome or amyotrophic lateral sclerosis) or a history of dysphagia or aspiration.
* Subjects with previous or current diagnosis of Bell's paresis.
* Subjects with known bleeding disorders or subjects who are taking thrombolytics or anticoagulants.
* Subjects who are taking anticholinergics or aminoglycoside antibiotics.
* Any prior surgery in the facial area that, in the opinion of the investigator, may interfere with the results.
* Subjects treated with fillers, HA filler or permanent filler, in the upper face one year or less from screening.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Assessment of severity of glabellar lines at rest and at maximum frown using the Merz Aesthetic 5-point scale. (However no primary outcome measure is defined in the study protocol) | Month 1
  To evaluate effect on glabellar line severity

OTHER OUTCOMES:
Assessment of severity of glabellar lines at rest and at maximum frown using the Merz Aesthetic 5-point scale | Day 0, 1, 3, 7, 14, month 3, 4 and 6
  To evaluate effect on glabellar line severity
Adverse Event reporting | Day 0-180
  To evaluate long term safety throughout the study period
Compound Muscle Action Potential (CMAP) reduction as percent of baseline CMAP measurement | Day 0, 1, 3, 7, month 1, 3 and 6
  To evaluate the Compound Muscle Action Potential using electroneurography

CONTACTS AND LOCATIONS:
Overall Officials: Anna Rostedt Punga, MD, Principal Investigator — ANNA Neuromuskulär Konsult
Locations (2):
- Sweden (2):
  - Göteborgs Plastikkirurgiska Center, Gothenburg
  - Anna Neuromuskulär Konsult, Uppsala